CLINICAL TRIAL: NCT00387426
Title: A Phase II Study of Sunitinib Malate in Idiopathic Myelofibrosis
Brief Title: Sunitinib in Treating Patients With Idiopathic Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00207; NCI-2009-00207 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000504056; 2006-0208; 2006-0208 (Other: M D Anderson Cancer Center); 7700 (Other: CTEP); N01CM62202 (NIH)
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2013-10

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Acute Undifferentiated Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Blastic Phase Chronic Myelogenous Leukemia; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Mast Cell Leukemia; Meningeal Chronic Myelogenous Leukemia; Primary Myelofibrosis; Progressive Hairy Cell Leukemia, Initial Treatment; Prolymphocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia; T-cell Large Granular Lymphocyte Leukemia; Untreated Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Myeloid Leukemia; Untreated Hairy Cell Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Mast-Cell; Primary Myelofibrosis; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic | interventions — Sunitinib

ARMS (1):
- Arm I (Experimental): Patients receive oral sunitinib malate once daily for 6 weeks.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate — Given PO

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with idiopathic myelofibrosis. Sunitinib may stop the growth of abnormal cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the abnormal cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the response rate and the duration of response in patients with idiopathic myelofibrosis treated with sunitinib malate.

SECONDARY OBJECTIVE:

I. Assess the safety of sunitinib malate in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral sunitinib malate once daily for 6 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks.

ELIGIBILITY:
Criteria:

* At least 4 weeks since prior chemotherapy or radiotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 4 weeks since prior major surgery
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including azole antifungals (ketoconazole and itraconazole), clarithromycin, erythromycin, diltiazem, verapamil, HIV protease inhibitors (indinavir, saquinavir, ritonavir, atazanavir, nelfinavir), and delavirdine
* At least 12 days since prior and no concurrent CYP3A4 inducers, including rifampin, rifabutin, carbamazepine, phenobarbital, phenytoin, Hypericum perforatum (St. John's wort), efavirenz, and tipranavir
* No prior antiangiogenic agents (e.g., bevacizumab, sorafenib, pazopanib, AZD2171, vatalanib, VEGF Trap)
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent therapeutic doses of coumarin-derivative anticoagulants (e.g., warfarin) (Warfarin =< 2 mg/day for prophylaxis of thrombosis and low molecular weight heparin allowed provided INR =< 1.5)
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent agents with proarrhythmic potential (e.g., terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, and flecainide)

Inclusion Criteria:

* Diagnosis of MF (histologically confirmed) requiring therapy, including those previously treated and relapsed or refractory (no more than one prior standard acute leukemia-type chemotherapy regimen; no limit on prior MF - directed therapies) or if newly diagnosed, with intermediate or high risk according to Lille scoring system (adverse prognostic factors are: Hb < 10 g/dl, WBC < 4 or > 30 x 10^9/L; risk group: 0 = low, 1 = intermediate, 2 = high), or with symptomatic organomegaly.
* Serum bilirubin levels </= 2x upper limit of the normal (ULN). Higher levels are acceptable if these can be attributed to active hemolysis or MF
* Serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels </= 2x ULN. Higher levels are acceptable if these can be attributed to MF.
* Serum creatinine levels </= 2x ULN.
* Eighteen years of age or older.
* ECOG performance status 0-1 (Karnofsky </= 70%).
* Patients must have QTc < 500 msec
* Women of childbearing potential and men must agree to use adequate contraception (e.g. hormonal or barrier method of birth control; abstinence) for the duration of study participation. All women of childbearing potential must have a negative pregnancy test prior to receiving sunitinib. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document
* Both men and women and members of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to beginning treatment or those who have not recovered from treatment-limiting adverse events (to grade 1 or better) due to agents administered more than 4 weeks earlier. At least 4 weeks must have elapsed since any major surgery prior to study enrollment. Continuous use of supportive care medications (i. e. growth factors, anagrelide, or hydroxyurea) is allowed.
* Patients may not be receiving any other investigational agents.
* Patients who have received prior treatment with any other specific antiangiogenic agent (e.g., bevacizumab, sorafenib, pazopanib, AZD2171, PTK787, VEGF Trap, etc.) targeting VEGF/VEGFR system. Other agents that may have some antiangiogenic effects are allowed). (i.e. thalidomide)
* Patients with abnormal QTc prolongation (defined as a QTc interval equal to or greater than 500 msec) or patients who have a history of serious ventricular arrhythmia (VT or VF>/= 3 beats in a row or other significant (as judged by treating physician) ECG abnormalities.Patients with consistently poorly controlled (during the month prior to study screening) hypertension (systolic blood pressure of 140 mmHg or higher or diastolic blood pressure of 90 mmHg or higher) despite appropriate medical management of the hypertension.
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin. Exceptions include: patients using warfarin of up to 2 mg daily for prophylaxis of thrombosis, and patients using low molecular weight heparin provided the patient's INR is </= 1.5.
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib tablets.
* Patients with any of the following conditions:·Serious or non-healing wound, ulcer, or bone fracture, history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment,·cerebrovascular accident (CVA) or transient ischemic attack, myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting, or pulmonary embolism within 12 months prior to study,·Class III or IV heart failure as defined by the NYHA functional classification system.
* Because sunitinib is metabolized primarily by the CYP3A4 liver enzyme, the eligibility of patients taking medications that are potent inducers or inhibitors of that enzyme will be determined following a review of their case by the Principal Investigator. Every effort should be made to switch patients taking such agents or substances to other medications.
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medications.
* Patients with uncontrolled intercurrent illness (as judged by treating physician) including, but not limited to, ongoing or active infections requiring IV antibiotics.
* Pregnant women are excluded from this study because sunitinib is an antiangiogenic agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sunitinib, breastfeeding should be discontinued if the mother is treated with sunitinib malate.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with sunitinib. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srdan Verstovsek, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 14, 2006 to December 17, 2007. All recruitment done at UT MD Anderson Cancer Center.
Groups:
- Sunitinib: 37.5 mg orally daily for 6-week cycle
Period: Overall Study
Arm/Group | Sunitinib
Started | 14
Completed | 0
Not Completed | 14
Not completed — Lack of Response | 7
Not completed — Toxicities | 4
Not completed — Disease Progression | 3

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 64 [51 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Clinical Response to Sunitinib Therapy
Description: Participant response assessed after two cycles of therapy according to categories: 1) complete response, 2) partial response, 3) clinical improvement, 4) stable disease 5) progressive disease, 6) early death from malignant disease, 7) early death from toxicity, 8) early death because of other cause, or 9) unknown (not assessable, insufficient data).
Time Frame: After two 6-week treatment courses (12 weeks)
Population: All participants assessed for response.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 14
participants | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 7/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=14)
Nausea (Gastrointestinal disorders) | 1 (2)
Optic Disc Edema (Blood and lymphatic system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pain (General disorders) | 1 (4)
Thrombosis Embolism (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 2 (2)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=14)
Nausea (Gastrointestinal disorders) | 5 (5)
Fatigue (General disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4)
High Blood Pressure (Cardiac disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Mucositis (Gastrointestinal disorders) | 1 (1)
Elevated Liver Function Tests (Metabolism and nutrition disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 9 (9)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 12 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less